CLINICAL TRIAL: NCT06999070
Title: A Randomized, Comparative Study of Different Doses of Intravenous Dexamethasone for Management of Post Spinal Anesthesia Shivering in Lower Limb Orthopedic Surgeries
Brief Title: The Effect of Different Doses of Dexamethasone on Post Spinal Anesthesia Shivering
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nader Ahmed Ahmed, A randomized, comparative study of different doses of intravenous dexamethasone for management of post spinal anesthesia shivering in lower limb orthopedic surgeries, Assiut University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: Dexamethasone and shivering
Record Dates: First submitted 2025-05-05; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Post Spinal Anesthesia Shivering
Keywords: Dexamethasone; Post spinal anesthesia shivering
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): Patients will take 0.1 mg/kg dexamethasone iv on incidence of Shivering after spinal anaethesia
  Interventions: Drug: Dexamethasone 0.1mg/kg
- Group B (Active Comparator): patients will take Dexamethasone 0.3 mg/kg intravenously injected to the patients after the detection of shivering
  Interventions: Drug: Dexamethasone 0.3mg/kg

INTERVENTIONS:
Drug: Dexamethasone 0.1mg/kg — On incidence of Shivering after spinal anaethesia
  Arms: Group A
Drug: Dexamethasone 0.3mg/kg — On incidence of Shivering after spinal anaethesia
  Arms: Group B

SUMMARY:
The precise etiology of post-spinal anesthesia shivering (PSAS) is not fully understood. The incidence ranges between 20 to 80%. Heat loss, reduced sympathetic tone and pyrogen release are termed as the main causes of intra/postoperative shivering.

The redistribution of heat from the core to the periphery of the body is facilitated by the vasodilatation associated with neuraxial anesthesia. Shivering causes tachycardia, lactic acidosis, hyperalgesia at the site of surgery, releases catecholamines, increases oxygen demand, and increases the risk of hypoxemia. [1][3] The most common causes of shivering include fever, shivering with spinal anesthesia movement disorders, post-anesthetic shivering, fear, excitement, stress, tremors, low blood sugar, anxiety, and shivering. Shivering with spinal anesthesia is an involuntary, oscillatory muscular activity that significantly increases metabolic heat production, potentially reaching up to 600% above the basal metabolic level.

Post-spinal shivering is one of the main sources of discomfort for patients recovering from surgery. Furthermore, it worsens wound pain and impedes electrocardiographic monitoring.

Prophylactic intravenous administration of dexamethasone has been currently used for controlling intra-operative and post spinal anesthesia shivering. Dexamethasone's anti-inflammatory effects may thereby lessen post-anesthesia shivering by reducing the gradient between skin and core body temperatures.

DETAILED DESCRIPTION:
Preoperative preparation:

All patients will be assessed preoperatively by history, physical examination, basal laboratory investigations (complete blood picture and INR) and electrocardiography (ECG). The anesthetic procedure will be explained to the patients and written informed consent will be signed. Preoperative preparations included fasting for 68 h before the surgery. No premedication was given to the patients prior to the surgery. On arrival of the patient in the operating room, heart rate, systolic blood pressure, diastolic blood pressure and mean arterial pressure (MAP), peripheral oxygen saturation (SpO2) and temperature will be recorded. A peripheral IV access will be obtained using an 18G venous cannula. IV fluids of normal room temperature will be given. No other warming device will be used. Lactated Ringers infused at 10 mL/kg/h over 30 min just before spinal anesthesia is administered. The infusion rate will be given as need till the end of surgery. Spinal anesthesia will be instituted at L34 or L 45 with patient in setting position with 2.5-4 mL (12.5-20 mg) of bupivacaine (heavy) 0.5% using a 25G Quinckes spinal needle. The level of sensory block will be assessed after intrathecal injection after 15 minutes.

Intraoperative management:

Standard (ASA) monitoring will be applied before anesthesia and monitored throughout the operation time Treatment of complications if occurred as: hypotension (defined as any decrease in mean arterial blood pressure (MAP) below 20% of the baseline or systolic pressure less than 90 mmHg) will be treated with a bolus of ephedrine (6-12 mg) I.V. Bradycardia (defined as decreased heart rate (HR) ≥ 20% compared to the baseline values) will be treated with 0.1 mg/kg IV atropine. Failed block or inadequate block (patient complains of pain in the intraoperative period), he/she will be given general anesthesia and will be excluded from the study.

The incidence and onset of PSAS were recorded, and Bedside Shivering Assessment Scale (BSAS) was used to grade the severity:

Grade 1 (zero points): No shivering Grade 2 (1 point): mild shivering that is limited to the neck and thorax may not be detected and may only be detected by palpation or as an artefact on ECG Grade 3 (2 points): Moderate: Intermittent upper extremity involvement plus/minus thorax Grade 4 (3 points): Severe: prolonged trembling of the upper or lower extremities or widespread shivering.

-The drug will be intravenously injected to the patients after the detection of shivering : Group A will take Dexamethasone 0.1 mg/kg Group B will take Dexamethasone 0.3 mg/kg. Monitoring the effect of the drug on shivering offset.

Postoperative Treatments:

At the end of the surgery, the patients will be transferred to the PACU. Patients will be kept in 45°C setting. Follow up the patient for 60 minutes (HR, SO2, BP and PSAS).

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II.
* Both sexes.
* Age: 21-55 years old.
* Scheduled for lower limb orthopedic surgery.
* BMI less than 35 kg/m2.

Exclusion Criteria:

* ASA physical status more than II.
* History of corticosteroid therapy or allergic reaction to any of the medication used in the study
* Patients with cognitive impairment.
* Pregnancy.
* Basal body temperatures of more than 38° or less than 36° C.
* BMI more than 35 kg/m2.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
severity of PSAS | 60 minutes after operation
  Bedside Shivering Assessment Scale (BSAS) was used to grade the severity:
  Grade 1 (zero points): No shivering Grade 2 (1 point): mild shivering that is limited to the neck and thorax may not be detected and may only be detected by palpation or as an artefact on ECG Grade 3 (2 points): Moderate: Intermittent upper extremity involvement plus/minus thorax Grade 4 (3 points): Severe: prolonged trembling of the upper or lower extremities or widespread shivering.

REFERENCES:
- See also: Mohamed Medhat Moustafa Kamal Nouh, Galal Adel Mohamed Abd Elrehiem Elkadi, Eman Mohamed Kamal Aboseif, Fasil Said Abd El Hamid, Marwa Mostafa Mohamed Ali Mowafi. A randomized, comparative study of prophylactic intravenous acetaminophen, dexamethasone an — https://www.apicareonline.com/index.php/APIC/article/view/2182/3323
- See also: Adel Rizk Botros, Yasser M. Nasr, Wafaa Ibrahim Abd el Wahid Khalil. Comparative study between dexamethasone and ondansetron for prevention ofshivering during spinal anaethesia. — https://zumj.journals.ekb.eg/article_56103_b019a045c46b4d6a524c9c617d742e10.pdf
- See also: Hunde Amsalu, Abebayehu Zemedkun, Teshome Ragasa, Yayeh Adamu. Evidence-Based Guideline on Prevention and Management of Shivering After Spinal Anesthesia in Resource-Limited Seettings — https://pubmed.ncbi.nlm.nih.gov/36090703/